CLINICAL TRIAL: NCT06231810
Title: Tracking a Tactile Signal Along the Nervous System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Netta Gurari, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-1256
Record Dates: First submitted 2024-01-08; First posted 2024-01-30 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Tactile Perception
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stimulus magnitude (Experimental): Differing levels of tactile stimulus will be applied
  Interventions: Behavioral: Tactile stimulation

INTERVENTIONS:
Behavioral: Tactile stimulation — Tactile stimuli of differing magnitudes will be applied

SUMMARY:
Quantify the flow of a tactile signal from the stimulus at the finger at the peripheral nervous system (PNS), to the central nervous system (CNS), and to cognitive perception at the brain in young adults (Aim 1) and individuals with and without stroke (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

-right-hand dominance for participants who are neurotypical

For Aim 1:

-age range of 18-23

For Aim 2:

* participants who are neurotypical will be a similar age to the participants with stroke
* participants who are neurotypical will have no musculoskeletal and neurological conditions
* participants with stroke will have a single stroke incident resulting in a unilateral lesion (ischemic and hemorrhagic)
* participants with stroke will be in the chronic phase (>1 year from stroke onset)
* participants with stroke will have an onset of stroke after the age of 18
* participants with stroke who meet the criteria of having the capacity to provide informed consent, regardless of aphasia

Exclusion Criteria:

* minors
* pregnant women
* prisoners
* adults not capable of consenting on their own behalf.

For Aim 2:

* participants with stroke who have used antispastic injections in the past six months
* participants with stroke who have a lesion in the brainstem and/or cerebellum
* participants with stroke who have a stroke arising due to brain surgery
* participants with stroke who have hemineglect

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Conscious detection threshold | 30 minutes during the first session of a one session protocol
  The magnitude at which a force stimulus applied to the finger can be first consciously detected. Different force levels will be applied, and the participant will indicate which of these forces can be detected. The changes in force applied will be in the units of N.

SECONDARY OUTCOMES:
Brain activation | 60 minutes during the first session of a one session protocol
  The magnitude and regions of brain activated in response to differing levels of force stimuli will be captured using fMRI. The % signal change in the brain will be used to define the brain activation in response to each force stimulus level.

OTHER OUTCOMES:
Peripheral nerve function | 30 minutes during the first session of a one session evaluation protocol
  Electrotactile stimuli will be applied to a finger, with the current (A) changing in magnitude. We will measure the level to which the peripheral nerve is activated using surface electrodes, which identify changes in voltage along the nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Netta Gurari, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No